CLINICAL TRIAL: NCT06622642
Title: Efficacy of Transoral Versus Transbuccal Technique for Fixation of Mandibular Angle Fracture in Terms of Mouth Opening and Radiographic Gap and Displacement
Brief Title: Efficacy of Transoral Versus Transbuccal Technique for Fixation of Mandibular Angle Fracture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Shanza Rehman, OMFS Resident, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1313-5995
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Mandibular Angle Fracture; Surgical Approach & Incisions
Keywords: Mandible trauma; Mandible angle fracture; Intraoral approach; Transbuccal approach; champy's prinicple of plating
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A will undergo transoral technique for mandibular angle fracture reduction (Active Comparator): In Group A transoral approach inferior alveolar nerve block and buccal nerve block will be given by 2% xylocaine with 1:100000 adrenaline. Incision will be made with surgical blade no 15 from gingival crevices of molars to ascending ramus. Fracture segments will be reduced alongwith MMF. A 5-hole 2mm miniplate with 2 holes anterior and 2 holes posterior to fracture line will be screwed to external oblique ridge and MMF will be removed and incision line will be closed
  Interventions: Procedure: Transoral technique for mandibular angle fracture reduction
- Group B will undergo transbuccal technique for mandibular angle fracture reduction (Experimental): In Group B tranbuccal technique approach inferior alveolar nerve block and buccal nerve block will be given by 2% xylocaine with 1:100000 adrenaline. Incision will be made with surgical blade no 15 from gingival crevices of molars to ascending ramus. Fracture segments will be reduced alongwith MMF after which extraorally a stab incision will be made with scalpel blade parallel to relaxed resting skin tension lines through which the cannula with a trocar will be inserted through facial tissue down to bone. Transbuccal instrument system will cionsist of transbuccal guide, mountable retractor, drill sleeve, drill guide, and 2mm drill bit. A 2mm titanium miniplate will be placed along buccal cortex and screwed through trocar system. MMF will be removed and incision line closed
  Interventions: Procedure: Transbuccal technique for mandibular angle fracture reduction

INTERVENTIONS:
Procedure: Transoral technique for mandibular angle fracture reduction — In transoral technique approach inferior alveolar nerve block and buccal nerve block will be given by 2% xylocaine with 1:100000 adrenaline. Incision will be made with surgical blade no 15 from gingival crevices of molars to ascending ramus. Fracture segments will be reduced alongwith MMF. A 5-hole 2mm miniplate with 2 holes anterior and 2 holes posterior to fracture line will be screwed to external oblique ridge and MMF will be removed and incision line will be closed.
  Arms: Group A will undergo transoral technique for mandibular angle fracture reduction
Procedure: Transbuccal technique for mandibular angle fracture reduction — In transbuccal technique inferior alveolar nerve block and buccal nerve block will be given by 2% xylocaine with 1:100000 adrenaline. Incision will be made with surgical blade no 15 from gingival crevices of molars to ascending ramus. Fracture segments will be reduced alongwith MMF. extraorally a stab incision will be made with scalpel blade parallel to relaxed resting skin tension lines through which the cannula with a trocar will be inserted through facial tissue down to bone. Transbuccal instrument system will cionsist of transbuccal guide, mountable retractor, drill sleeve, drill guide, and 2mm drill bit. A 2mm titanium miniplate will be placed along buccal cortex and screwed through trocar system. MMF will be removed and incision line closed
  Arms: Group B will undergo transbuccal technique for mandibular angle fracture reduction

SUMMARY:
The goal of this clinical trial is to learn if transbuccal technique for mandibular angle fracture is better than transoral technique. The main questions it aims to answer are:

* Does transbuccal technique provide better mouth opening than transoral technique
* Radiographic gap and displacement between fracture lines is more prevalent in transoral technique than transbuccal technique postoperatively Researcher will compare both the techniques to see if transbuccal technique works better than transoral technique

Participants will:

* Be assessed 1 week , 1 month and 3 months postoperatively
* Their mouth opening will be assessed by measuring interincisal opening with ruler
* Radiographic gap between fracture segments and displacement of fractured segments will be measured on OPG through ruler

DETAILED DESCRIPTION:
OBJECTIVE: To compare the efficacy of transoral versus transbuccal technique for fixation of mandibular angle fracture in terms of mouth opening and radiographic gap and displacement.

OPERATIONAL DEFINITIONS:

MANDIBLE ANGLE FRACTURE:Fracture line in area bound from the anterior border of the masetter(distal of 2nd molar) to posterior border of the masetter assessed clinically through palpation and radiographically through OPG and PA mandible.

EFFICACY: The efficacy of the two procedures will be assessed on 1 week, 1 month, 3 months with following outcomes.

1. MOUTH OPENING: Mouth opening will be defined as maximum interincisal distance measured in millimeters through ruler.
2. GAP BETWEEN FRACTURE SEGMENTS: Gap between proximal and distal fracture lines measured in millimeters in OPG with ruler.
3. DISPLACEMENT OF FRACTURE SEGMENTS: Presence of step between distal and proximal segments in vertical plane at the lower border on OPG.

HYPOTHESIS: Transbuccal approach will have better functional post-operative mouth opening, radiographic gap and displacement compared to transoral fixation technique in patients with mandibular angle fracture.

MATERIALS AND METHODS:

STUDY DESIGN: Prospective randomized clinical study. SETTING:Oral and maxillofacial surgery department, emergency and OPD of Services Hospital Lahore.

DURATION OF STUDY: Six months after approval of synopsis. SAMPLE SIZE: Sample size was calculated through openepi calculator for sample size for % frequency in a population(random sample) Population size=1000000 Anticipated % frequency(p)=50 Confidence limits=12% absolute precision Design effect=1.0 for random sample Sample size for 95% confidence level=67 Sample size in each group=n=34

SAMPLING TECHNIQUE: Nonprobability purposive sampling technique.

SAMPLE SELECTION:

DATA COLLECTION PROCEDURE:

METHODS OF DATA COLLECTION:Patients fulfilling inclusion criteria will be taken from emergency and OPD of Services Hospital Lahore and will be randomized into 2 groups group A( transoral technique) and group B (transbuccal technique) by lottery method after taking informed consent from them by briefing them about study, research protocol and risk-benefit ratio.Diagnosis and treatment plan will be made based on history, clinical examination and radiographic findings of OPG and PA mandible. Procedure will be done by single surgical team. In Group A transoral approach inferior alveolar nerve block and buccal nerve block will be given by 2% xylocaine with 1:100000 adrenaline. Incision will be made with surgical blade no 15 from gingival crevices of molars to ascending ramus. Fracture segments will be reduced alongwith MMF. A 5-hole 2mm miniplate with 2 holes anterior and 2 holes posterior to fracture line will be screwed to external oblique ridge and MMF will be removed and incision line will be closed. In Group B tranbuccal technique same procedure will be performed till fracture reduction and MMF after which extraorally a stab incision will be made with scalpel blade parallel to relaxed resting skin tension lines through which the cannula with a trocar will be inserted through facial tissue down to bone. Transbuccal instrument system will cionsist of transbuccal guide, mountable retractor, drill sleeve, drill guide, and 2mm drill bit. A 2mm titanium miniplate will be placed along buccal cortex and screwed through trocar system. MMF will be removed and incision line closed.

DATA COLLECTION TOOLS:All study variables will be assessed by single person at 1 week,1 month and 3 months post op.Clinical parameters will be assessed through proforma/questionnaire. Radiological parameters will be assessed through OPG, PA mandible.

DATA ANALYSIS PROCEDURE:Data will be collected and statistically analyzed using the SPSS software version 29. Mean and standard deviation will be calculated for quantitative variables like age, etiology, associated fractures, clinical and radiological parameters. Frequency and percentage will be measured for qualitative measures like gender, site. Efficacy between both groups will be compared by t-test and a P value of less than or equal to 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1.All dentate and partially dentate patients with unilateral mandibular angle fracture.
* 2. Both isolated mandibular angle fractures and mandibular angle fractures associated with other facial fractures will be included

Exclusion Criteria:

* 1.Comminuted mandibular angle fractures.
* 2.Edentulous patients.
* 3. Gross external laceration in submandibular region.
* 4.Presence of local bone pathology alongwith fracture will be excluded from study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean of mouth opening | 1 week, 1 month, 3 month
  Mouth opening will be defined as maximum interincisal distance measured in millimeters through ruler.
MEAN OF GAP BETWEEN FRACTURE SEGMENTS | 1 week, 1 month, 3 month
  Gap between proximal and distal fracture lines measured in millimeters in OPG with ruler.
MEAN OF DISPLACEMENT OF FRACTURE SEGMENTS: | 1 week, 1 month, 3 month
  Presence of step between distal and proximal segments in vertical plane at the lower border on OPG.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 9. Hidayatullah SK, Saifullah SK. Outcome of Transbuccal and Transoral Technique in Open Reduction and Internal Fixation of Mandibular Angle Fractures. Pak J Med Health Sci. 2022 Jul 30;16(07):85-85
- [Background] 8. Elsayed SA, Reda HM, Awadd MM, Mourad SI, Shokeir HM, Elsayed EH, Al-Moraissi. Transbuccal vs intraoral approach using an angulated screwdriver in fixation of a mandibular angle fracture. Open Dent J. 2022 Aug 16(1):1-7
- [Background] 7. Gupta S, Pandilwar P, Yerragudi N, Chawla JG, Redij S, Kumbhare S. Fixation of mandibular angle fracture by transoral approach versus transbuccal approach a clinical .and radiographic study.Asian J Contemp Dent Sci.2021 March 1(1):04-07
- [Background] 6. Asim M,Muddassar M,Qureshi IS,Rana ZA, Hoti KK. Comparison of intraoral external oblique ridge fixation and transbuccal lateral cortical plate fixation for mandibular angle fracture-A randomized control trial. Health Sci J. 2020;14(3):716.
- [Background] Sehrawat K, Malik B, Vallabha HV, Vaishnavi AB, Pendyala SK, Ibrahim M, Binyahya FA. A Comparative Evaluation of Transbuccal versus Transoral Approach for the Management of Mandibular Angle Fractures: A Prospective, Clinical, and Radiographic Study. J Pharm Bioallied Sci. 2021 Nov;13(Suppl 2):S1295-S1299. doi: 10.4103/jpbs.jpbs_112_21. Epub 2021 Nov 10. PMID 35017974
- [Background] Bhardwaj B, Singh J, Mahajan S. Transbuccal Approach in Management of Mandible Angle Fracture. Indian J Otolaryngol Head Neck Surg. 2020 Dec;72(4):457-462. doi: 10.1007/s12070-020-01904-y. Epub 2020 Jun 23. PMID 33088775
- [Background] Krishnan Kutty D, Hallur N, Siddiqa A, Zakaullah S, Kothari C. Management of Sub-Condylar and Angle of Mandible Fracture by a Trans-Buccal Trocar Along With an Intra-Oral Approach. Indian J Otolaryngol Head Neck Surg. 2020 Dec;72(4):538-544. doi: 10.1007/s12070-020-02058-7. Epub 2020 Aug 20. PMID 33088789
- [Background] 2. Khokhar M, Sadhwan BS, Tailor SS. Comparison of intra-oral and extra-oral approaches in mandibular angle fractures. Nat J Clinic Orthop 2022; 6(3): 01-03
- [Background] Pavithra SK, Vivek N, Saravanan C, Karthik R, Prashanthi G, Scott C. Comparison of Conventional Versus Right Angled Fixation Technique in Management of Mandibular Angle Fractures - A Prospective Randomized Clinical Study. J Oral Maxillofac Surg. 2023 Aug;81(8):1001-1010. doi: 10.1016/j.joms.2023.04.005. Epub 2023 Apr 20. PMID 37160255